CLINICAL TRIAL: NCT03233581
Title: Improving Physical Activity in Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Jason Mendoza, Investigator and Associate Professor of Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fitbit YA 9865
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Physical Activity; Quality of Life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitbit + Facebook + Health Coaching (Experimental): Participants will use the Fitbit device and join the Facebook group. They will also receive brief weekly health coaching from a research staff. Participants will select an adult family member or friend to also receive a Fitbit during the intervention period to provide them with support.
  Interventions: Behavioral: Fitbit + Facebook + Coaching Group
- Usual care control with Fitbit only (Active Comparator): Participants will be loaned a Fitbit device only. They will not join the Facebook group nor receive health coaching. They will not select an adult family member or friend to receive a Fitbit device to provide them with support.
  Interventions: Behavioral: Fitbit only

INTERVENTIONS:
Behavioral: Fitbit + Facebook + Coaching Group — Participants will use the FitBit device to track their physical activity (PA). Participants will receive and post messages and receive badges on the Facebook group. Weekly a research staff member will call them to provide brief health coaching. Participants will select an adult family member or friend to also receive a Fitbit during the intervention period to provide support.
  Arms: Fitbit + Facebook + Health Coaching
Behavioral: Fitbit only — Participants will receive a Fitbit device only, and will not receive health coaching, join the Facebook group, or select an adult family member or friend to receive a Fitbit to provide them with support.
  Arms: Usual care control with Fitbit only

SUMMARY:
The Primary Goal is to conduct a 12 week pilot randomized controlled trial (RCT) of the Fitbit Flex, a popular, affordable, wearable physical activity tracking device, and the Fitbit mobile health (mHealth) app. The target population will be cancer survivors 18-39 years old recruited from the Seattle Cancer Care Alliance. For the intervention group, peer influences will be engaged via a private, social network (e.g. a Facebook group) customized for survivors. Measurements will be completed (1) at baseline, prior to randomization, and (2) during the final week of the intervention period (follow-up measure). This pilot study will provide initial proof of concept and allow for further customization of the intervention for cancer survivors in anticipation of a future, larger proposal to study physical activity and related outcomes over a multi-year period.

Besides conducting exploratory analyses of primary and secondary outcomes for this pilot RCT, we also specify feasibility criteria including: (1) recruiting 50 cancer survivors ages 18-39 years and between 1.0-5.0 years from the completion of active cancer therapy, (2) intervention participants wear the Fitbit Flex on the majority of all intervention days during the 12-week intervention period, and (3) ≥75% of all participants complete online questionnaire data collection at Time 1 and Time 2.

ELIGIBILITY:
Inclusion Criteria:

* Does not meet recommended guidelines for physical activity (PA,150 min of moderate activity or 75 min of vigorous activity)
* Currently between 1.0-5.0 years from the completion of active cancer therapy
* Able to read and speak English
* Have a smart phone (or can borrow a study-provided iPod Touch) and willing to use it for the mobile app and Facebook group

Exclusion Criteria:

* Pregnant or planning on becoming pregnant in the next year

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-05-06 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Post-intervention physical activity (minutes per day of moderate-to-vigorous physical activity objectively measured by accelerometers) | up to week 12

SECONDARY OUTCOMES:
Post-intervention health related quality of life (measured by questionnaire) | up to week 12
Self-determination theory constructs (measured by the Behavioral Regulation in Exercise Questionnaire 2) | up to week 12

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Children's Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson AM, Baker KS, Haviland MJ, Syrjala KL, Abbey-Lambertz M, Chow EJ, Mendoza JA. A Pilot Randomized Controlled Trial of a Fitbit- and Facebook-Based Physical Activity Intervention for Young Adult Cancer Survivors. J Adolesc Young Adult Oncol. 2022 Aug;11(4):379-388. doi: 10.1089/jayao.2021.0056. Epub 2021 Oct 22. PMID 34677081
- [Derived] Miropolsky EM, Scott Baker K, Abbey-Lambertz M, Syrjala K, Chow EJ, Ceballos R, Mendoza JA. Participant Perceptions on a Fitbit and Facebook Intervention for Young Adult Cancer Survivors: A Qualitative Study. J Adolesc Young Adult Oncol. 2020 Jun;9(3):410-417. doi: 10.1089/jayao.2019.0072. Epub 2020 Jan 13. PMID 31928489